CLINICAL TRIAL: NCT04424836
Title: the Effect of HFNC Treatment on Mortality and Length of ICU Stay in Patient With COVID-19 Pneumonia
Brief Title: HFNC Treatment in COVID-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Altınay, specialist medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 5569
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus Infection; Pneumonia, Viral; Acute Respiratory Failure
Keywords: high flow nasal cannula (HFNC); conventional oxygen treatment (COT)
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- H GROUP: patients get the oxygen supply with high flow nasal cannula . In group H, HFNC device settings the initial flow rate was 30 L/min and could be increased to 60. The Fio2 was adjusted to maintain oxygen saturation as indicated by a pulse oximetry reading of grater than or equal to %90.
  Interventions: Device: high flow nasal cannula device
- C GROUP: patients get the oxygen supply with conventional methods. In group C 6-15 L/min oxygen delivered to patients by conventional methods and targeted to maintain the oxygen saturation %90 or over.

INTERVENTIONS:
Device: high flow nasal cannula device — device is supplying oxygen with heated and humidified air in a high flow rate
  Groups: H GROUP

SUMMARY:
coronavirus disease 2019 related pneumonia is causing acute respiratory failure and this is the most common reason for ICU admission. We have several different way for respiratory support. HFNC is one of the new technics for oxygen support. Our main purpose to observe the effect of HFNC on coronavirus disease 2019 patients' ICU stay and mortality.

DETAILED DESCRIPTION:
In the first group (group H), the data of patients undergoing HFNC treatment, and in group II (Group K), the data of patients who received COT with a reservoir mask were included.

In HFNC support, the current air temperature is 31-37 degrees, the flow rate is 30-60 lt / min, and the FiO2 value is targeted so that saturation is 93% and above. Initially, continuous treatment was applied intermittently after the partial oxygen pressure / fraction of inspired oxygen(fio2) ratio exceeded 250 and clinical well-being occurred.

In patients in Group K, fingertip saturation was targeted as 93% and above, and a COT was applied with a reservoir mask with a flow rate of 6-15 l / min.

The flow rate was calculated using the formula of FiO2 (%) = 21 + 4 * (liters / min) in patients undergoing COT. Noninvasive mechanical ventilation was applied to patients who could not be provided with adequate clinical and laboratory well-being in both groups (partial oxygen pressure / fraction of inspired oxygen ratio below 150) and invasive mechanical ventilation if this was insufficient.

ELIGIBILITY:
Inclusion Criteria:

* We include the patient with acute respiratory failure related coronavirus disease 2019 (diagnosed with polymerase Chain Reaction), older than 18 year and supported by High Flow Nasal cannulae or conventional oxygen treatment(COT).

Exclusion Criteria:

* Patients with primary pulmonary disease, Glasgow Coma scale≤ 12 , respiratory acidosis in the first blood gases(ph≤ 7,2 - pCO2≥50) will exclude.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: coronavirus disease 2019 patients admitted to the ICU for acute respiratory failure 15 march to 15 may
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
short term mortality | in 28 days.
  the mortality rate of patients
icu stay | up to 28 days
  means the stay day of patients in intensive care unit

SECONDARY OUTCOMES:
blood gases | at the admission time and 24th hour
  partial oxygen pressure, partial carbon dioxide pressure . both measured in mmhg

CONTACTS AND LOCATIONS:
Overall Officials: ayse su cinar, Study Chair
Locations (1):
- Sisli Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Result] Arabi YM, Arifi AA, Balkhy HH, Najm H, Aldawood AS, Ghabashi A, Hawa H, Alothman A, Khaldi A, Al Raiy B. Clinical course and outcomes of critically ill patients with Middle East respiratory syndrome coronavirus infection. Ann Intern Med. 2014 Mar 18;160(6):389-97. doi: 10.7326/M13-2486. PMID 24474051
- [Result] Akerstrom S, Gunalan V, Keng CT, Tan YJ, Mirazimi A. Dual effect of nitric oxide on SARS-CoV replication: viral RNA production and palmitoylation of the S protein are affected. Virology. 2009 Dec 5;395(1):1-9. doi: 10.1016/j.virol.2009.09.007. Epub 2009 Oct 1. PMID 19800091

DOCUMENTS (2):
  • Study Protocol (2020-06-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT04424836/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT04424836/SAP_001.pdf